CLINICAL TRIAL: NCT01506323
Title: Portable Mantram Meditation for Veterans With Military Related PTSD
Brief Title: Mantram Repetition Meditation for Veterans With PTSD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPLE-003-11S
Record Dates: First submitted 2011-12-19; First posted 2012-01-10 (Estimated); Results first posted 2015-09-02 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Complementary Therapy; Stress Disorders, Post-Traumatic; Veterans Health; Clinical Trials, Randomized; Mindfulness; Spirituality; Meditation; Mind-body therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mantram Repetition Program (MRP) (Experimental): A portable meditation-based "Mantram Repetition Program (MRP)" will be delivered individually in 8-weekly 1 hour sessions to teach a set of strategies for training attention to manage symptoms. For this study, the program targets symptoms of posttraumatic stress disorder (PTSD) in Veterans who have experienced military-related trauma.
  Interventions: Behavioral: Mantram Repetition Program (MRP)
- Present Centered Therapy (PCT) (Active Comparator): Present Centered Therapy (PCT) is a form of individually-delivered 8-weekly, 1 hour sessions that are problem-oriented to improve current coping. For this study, it served as an attention control arm for the non-specific effects of individual therapist interaction.
  Interventions: Behavioral: Present Centered Therapy (PCT)

INTERVENTIONS:
Behavioral: Mantram Repetition Program (MRP) — The MRP teaches three portable, mindfulness strategies to train attention and manage symptoms: 1) Mantram (sacred word) Repetition, 2) Slowing Down, and 3) One-Pointed Attention. These tools are presented as working together synergistically and cumulatively, over time, to interrupt negative thoughts, behaviors, and emotional states such as anger, rage, irritability and impatience. Participants choose their own words or phrases and are encouraged to practice repeating a mantram at any time or place. In this study, MRP is delivered individually in eight weekly, 1-hour sessions, using a standardized manual, instructor guide, and homework assignments for experiential learning.
  Other Names: MRP, Mantram Meditation
  Arms: Mantram Repetition Program (MRP)
Behavioral: Present Centered Therapy (PCT) — The PCT is a form of individual therapy that is problem-oriented to improve current coping. It avoids details of traumatic experiences. In this study, it is delivered individually in 8 weekly, 1 hour sessions to serve as an active, attention control arm. Sessions are unstructured and managed so that there is some engagement of the participant's emotional concerns with an emphasis on strengths and process encouragement rather than skills training. Three components of PCT include 1) developing a therapeutic relationship for social support, 2) focusing on current problems and problem solving, 3) and setting goals.
  Other Names: PCT
  Arms: Present Centered Therapy (PCT)

SUMMARY:
The aim of this study was to determine the usefulness of a portable, meditation-based intervention called the Mantram Repetition Program (MRP) for Veterans with military-related posttraumatic stress disorder (PTSD). This study compared the individual delivery of the MRP to individual delivery of Present-Centered Therapy (PCT) at two sites in San Diego, California, and Bedford, Massachusetts.

DETAILED DESCRIPTION:
The investigators conducted a prospective, parallel group, two-site, randomized clinical trial on the therapeutic treatment efficacy of the Mantram Repetition Program (MRP) by offering it as a stand-alone intervention, compared to an attention control condition of Present Centered Therapy (PCT) in a diverse sample of Veterans with post-traumatic stress disorder (PTSD). Primary outcomes included clinician-assessed and self-reported PTSD symptom severity. Secondary outcomes included insomnia, depression, anger, spiritual well-being, and mindfulness. Veterans were were recruited from a variety of clinics, including primary care, women's health, and specialty clinics in two geographical locations within the Department of Veterans Affairs healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Read and write English fluently
* Traumatic event related to military-duty, including combat, military training accidents, and military sexual trauma
* Transportation to attend meetings and available to complete study protocols
* Stable dose and type of PTSD medications for at least 6 weeks (per chart review)
* Willing to track medication changes during study

Exclusion Criteria:

* Inability to give informed, voluntary consent
* Cognitive impairment sufficient to cause inability to complete the protocol
* Psychotic symptoms
* Dementia or other organic mental disorders that may cause inability to complete the protocol
* Significant documented alcohol/substance abuse
* Presence of severe suicidal urges or intent
* Residence in a geographical area outside of San Diego County or Bedford, Massachusetts area
* Current daily practice of any skills of any meditation-based program - including, but not limited to:

  * Transcendental Meditation (TM)
  * Yoga
  * Tai Chi
  * Qi-Gong
  * Vipassana or Insight Meditation
  * Loving-Kindness or Compassion Meditation
  * Mindfulness-Based Stress Reduction (MBSR) or other mindfulness program
  * Guided Imagery
  * Mantram Repetition
  * Passage Meditation
  * Walking Meditation
  * Zen or Buddhist meditation
  * Self-hypnosis, Bio-feedback, etc.
* Other participant circumstances that, in the opinion of a consensus of the study team, would interfere with the safety of prospective participants or their need for treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2012-01; Primary Completion 2014-03 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill E. Bormann, PhD RN, Principal Investigator — San Diego Veterans Healthcare System; A. Rani Elwy, PhD MSc BA, Principal Investigator — Edith Nourse Rogers Memorial Veterans Hospital
Locations (2):
- United States (2):
  - VA San Diego Healthcare System, San Diego, California
  - Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA, Bedford, Massachusetts

REFERENCES:
- [Result] Bormann JE, Plumb DN, Beck DJ, Glickman M, Zhao S, Osei-Bonsu PE, Johnston JM, Herz L, Elwy AR. Portable meditation-based mantram program reduces PTSD symptoms in veterans: A randomized controlled trial. Poster session presented at: International Society for Traumatic Stress Studies Annual Symposium; 2014 Nov 1; Miami, FL.
- [Derived] Malaktaris A, McLean CL, Mallavarapu S, Herbert MS, Kelsven S, Bormann JE, Lang AJ. Higher frequency of mantram repetition practice is associated with enhanced clinical benefits among United States Veterans with posttraumatic stress disorder. Eur J Psychotraumatol. 2022 Jun 10;13(1):2078564. doi: 10.1080/20008198.2022.2078564. eCollection 2022. PMID 35713599
- [Derived] Bormann JE, Thorp SR, Smith E, Glickman M, Beck D, Plumb D, Zhao S, Ackland PE, Rodgers CS, Heppner P, Herz LR, Elwy AR. Individual Treatment of Posttraumatic Stress Disorder Using Mantram Repetition: A Randomized Clinical Trial. Am J Psychiatry. 2018 Oct 1;175(10):979-988. doi: 10.1176/appi.ajp.2018.17060611. Epub 2018 Jun 20. PMID 29921143
- See also: Home Page: Dr. Jill E. Bormann — http://www.jillbormann.com
- See also: Bormann, JE presented VA Cyberseminar Presentation, February 2015. Symptom management for PTSD: Mantram Repetition Program randomized clinical trial results. — http://www.hsrd.research.va.gov/for_researchers/cyber_seminars/archives/video_archive.cfm?SessionID=928

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Veterans with a history of military-related posttraumatic stress disorder (PTSD) were recruited from January 2012 to March 2014 from outpatient clinics and primary care providers at the VA San Diego Healthcare System in San Diego, CA, and the Edith Nourse Rogers Memorial VA Hospital in Bedford, MA.
Pre-assignment Details: Five (5) enrolled participants were excluded from the trial before assignment to groups due to:
  1) lost to follow-up; 2) could not commit to the study; 3) transportation difficulties. Three (3) participants were missing significant demographic data, resulting in a total of 173 for the analysis.
Groups:
- Mantram Repetition Program (MRP): The MRP teaches three portable, mindfulness strategies to train attention and manage symptoms: 1) Mantram (sacred word) Repetition, 2) Slowing Down, and 3) One-Pointed Attention. These tools are presented as working together synergistically and cumulatively, over time, to interrupt negative thoughts, behaviors, and emotional states such as anger, rage, irritability and impatience. Participants choose their own words or phrases and are encouraged to practice repeating a mantram at any time or place. In this study, MRP was delivered individually in eight weekly, 1-hour sessions, using a standardized manual, instructor guide, and homework assignments for experiential learning.
- Present Centered Therapy (PCT): The PCT is a form of individual therapy that is problem-oriented to improve current coping. It typically avoids actual details of traumatic experiences. In this study, it is delivered individually in 8 weekly, 1 hour sessions to serve as an active, attention comparison arm. Sessions are unstructured and managed so that there is some engagement of the participant's emotional concerns with an emphasis on strengths and process encouragement rather than skills training.
Period: Overall Study
Arm/Group | Mantram Repetition Program (MRP) | Present Centered Therapy (PCT)
Started | 89 | 84
Post-treatment Completers | 69 | 72
Post-treatment Completed CAPS | 68 | 72
Completed | 65 | 71
Not Completed | 24 | 13
Not completed — Lost to Follow-up | 5 | 4
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Lack of Efficacy | 1 | 3
Not completed — Moved out of area | 5 | 2
Not completed — Schedule or Transportation conflict | 8 | 0
Not completed — Started another treatment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Mantram Repetition Program (MRP): The Mantram Repetition Program (MRP) teaches three portable, mindfulness strategies to train attention and manage symptoms: 1) Mantram (sacred word) Repetition, 2) Slowing Down, and 3) One-Pointed Attention. These tools are presented as working together synergistically and cumulatively, over time, to interrupt negative thoughts, behaviors, and emotional states such as anger, rage, irritability and impatience. Participants choose their own words or phrases and are encouraged to practice repeating a mantram at any time or place. In this study, MRP was delivered individually in eight weekly, 1-hour sessions, using a standardized manual, instructor guide, and homework assignments for experiential learning.
- Present Centered Therapy (PCT): Present Centered Individual Therapy (PCT): The PCT is a form of individual therapy that is problem-oriented to improve current coping. It avoids details of traumatic experiences. In this study, it is delivered individually in 8 weekly, 1 hour sessions to serve as an active, attention control arm. Sessions are unstructured and managed so that there is some engagement of the participant's emotional concerns with an emphasis on strengths and process encouragement rather than skills training.
- Total: Total of all reporting groups
Arm/Group | Mantram Repetition Program (MRP) | Present Centered Therapy (PCT) | Total
Number analyzed (Participants) | 89 | 84 | 173
Age, Categorical [Count of Participants; unit: Participants] — Baseline data was collected from participants who scored greater or equal to 50 on the PTSD Checklist-Military (PCL-M) and greater or equal to 45 on the Clinician Administered PTSD Scale (CAPS).
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 74 | 70 | 144
    >=65 years | 15 | 14 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 10 | 26
  Male | 73 | 74 | 147
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 17 | 30
  Not Hispanic or Latino | 76 | 67 | 143
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 4 | 6
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 14 | 11 | 25
  Black or African American | 1 | 6 | 7
  White | 60 | 51 | 111
  More than one race | 8 | 10 | 18
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 89 | 84 | 173

OUTCOME MEASURES:

1. Primary Outcome: Clinician-Administered PTSD Scale (CAPS) Diagnostic and Statistical Manual, 4th ed., Text Revision (DSM-IV)
Description: PTSD symptom severity is measured by CAPS to determine PTSD diagnosis. The scale rates 17 items representing the Diagnostic and Statistical Manual IV (DSM-IV) criteria B (re-experiencing), C (avoidance/numbing) and D (hyper-arousal). CAPS has demonstrated high levels of internal consistency, good inter-rater reliability, & excellent convergent validity. The F1/I2 rule will be applied to establish the diagnosis of PTSD aligned with DSM-IV (e.g. one symptom of Criterion B, three of Criterion C, and two of Criterion D. The CAPS also includes an item to assess duration of PTSD symptoms. CAPS total score ranges from 0-136 with higher scores indicating greater symptom severity.
Time Frame: Baseline to post-treatment (week 8); Baseline to 2 months post-treatment.
Population: Intent to treat analysis included 89 MRP and 84 PCT participants. Completers at post-treatment included 69 MRP and 72 PCT participants. Completers at 2-months follow up included 65 MRP and 71 PCT participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Present Centered Therapy (PCT): The PCT is a form of individual therapy that is problem-oriented to improve current coping. It typically details of traumatic experiences. In this study, it is delivered individually in 8 weekly, 1 hour sessions to serve as an active, attention comparison arm. Sessions are unstructured and managed so that there is some engagement of the participant's emotional concerns with an emphasis on strengths and process encouragement rather than skills training. Three components of PCT include 1) developing a therapeutic relationship for social support, 2) focusing on current problems and problem solving, 3) and setting goals.
Arm/Group | Mantram Repetition Program (MRP) | Present Centered Therapy (PCT)
Number analyzed (Participants) | 89 | 84
units on a scale
  Baseline | 77.46 (16.48) | 75.61 (16.83)
  Post-treatment | 52.39 (22.60) | 62.07 (23.42)
  2 months follow-up | 50.62 (23.21) | 59.00 (22.79)
Statistical Analysis 1: Comparison: Mantram Repetition Program (MRP) vs Present Centered Therapy (PCT); This analysis is from baseline (week 0) to post-treatment (week 8). Cronbach's alpha for this study was .92 at baseline; Test type: Superiority or Other; p < .006, Mixed Models Analysis — This p-value is based on a false discovery rate adjustment for multiple hypothesis testing; Mixed-effects, repeated measures models adjusting for demographic factors were implemented
Statistical Analysis 2: Comparison: Mantram Repetition Program (MRP) vs Present Centered Therapy (PCT); This analysis is from baseline (week 0) to 2 months follow-up; Test type: Superiority or Other; p < .031, Mixed Models Analysis — The p-value was adjusted for multiple comparisons using false discovery rate; This p-value is based on a false discovery rate adjustment for multiple hypothesis testing; repeated measures

2. Primary Outcome: Re-experiencing Subscale (Criterion B) on the Clinician Administered PTSD Scale (CAPS)
Description: This subscale measures the frequency and intensity of (1) recurrent or intrusive recollections of trauma, (2) recurrent, distressing dreams of the trauma, (3) acting as if the traumatic event were recurring like a flashback, (4) intense psychological distress at exposure to internal or external cues that resemble the trauma; and/or (5) physiological reactivity on exposure to internal or external cues that symbolize or resemble an aspect of the trauma. Duration of these symptoms is greater than one month and symptoms cause clinically significant distress or impairment in social, occupational, or other important areas of of functioning. Scores can range from 0 to 40 and higher scores mean greater severity of re-experiencing.
Time Frame: Baseline to post-treatment (week 8); Baseline to 2 months post-treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mantram Repetition Program (MRP) | Present Centered Therapy (PCT)
Number analyzed (Participants) | 89 | 84
units on a scale
  Baseline | 20.74 (7.63) | 21.80 (6.42)
  Post-treatment | 14.40 (8.71) | 15.78 (9.12)
  2-months follow-up | 14.32 (8.73) | 15.94 (8.99)
Statistical Analysis 1: Comparison: Mantram Repetition Program (MRP) vs Present Centered Therapy (PCT); This analysis is from baseline to post-treatment. Cronbach's alpha for this study was .86 at baseline; Test type: Superiority or Other; p = 0.82, Mixed Models Analysis — The p-value is based on false discovery rate adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Mantram Repetition Program (MRP) vs Present Centered Therapy (PCT); This analysis is from baseline to 2 months post-treatment; Test type: Superiority or Other; p = 0.82, Mixed Models Analysis — This p-value is based on a false discovery rate adjustment for multiple hypothesis testing

3. Primary Outcome: Avoidance Subscale (Criterion C) on the Clinician Administered PTSD Scale (CAPS)
Description: This subscale measures the frequency and intensity of persistent avoidance of stimuli associated with the trauma and numbing of general responsiveness as indicated by 3 or more of the following: (1) efforts to avoid thoughts, feelings, or conversations associated with the trauma, (2) efforts to avoid activities, places or people that arouse recollections of the trauma, (3) inability to recall an important aspect of the trauma, (4) markedly diminished interest or participation in significant activities, (5) feelings of detachment or estrangement from others, (6) restricted range of affect, and/or (7) sense of a foreshortened future. Duration of these symptoms is greater than one month and causes clinically significant distress or impairment in social, occupational, or other important areas of of functioning. Scores range from 0 to 56 with higher scores indicating greater severity of avoidance.
Time Frame: Baseline to post-treatment (week 8); Baseline to 2 months post-treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mantram Repetition Program (MRP) | Present Centered Therapy (PCT)
Number analyzed (Participants) | 87 | 81
units on a scale
  Baseline | 29.92 (8.29) | 29.13 (8.87)
  Post-treatment | 19.91 (10.50) | 24.13 (11.18)
  2-months follow-up | 18.67 (11.61) | 21.78 (10.90)
Statistical Analysis 1: Comparison: Mantram Repetition Program (MRP) vs Present Centered Therapy (PCT); This analysis is from baseline to post-treatment. Cronbach's alpha for this study was .85 at baseline; Test type: Superiority or Other; p < 0.008, repeated measures — This p-value is based on a false discovery rate adjustment for multiple hypothesis testing
Statistical Analysis 2: Comparison: Mantram Repetition Program (MRP) vs Present Centered Therapy (PCT); This analysis is from baseline to 2 months post-treatment; Test type: Superiority or Other; p < 0.09, Mixed Models Analysis — This p-value is based on a false discovery rate adjustment for multiple hypothesis testing

4. Primary Outcome: Hyperarousal (Criterion D) on the Clinician Administered PTSD Scale (CAPS)
Description: This subscale measures the frequency and intensity of increased arousal as indicated by two or more of the following: (1) difficulty falling or staying asleep, (2) irritability or outbursts of anger, (3) difficulty concentrating, (4) hypervigilance, and/or (5) exaggerated startle response. Duration of these symptoms is greater than one month and causes clinically significant distress or impairment in social, occupational, or other important areas of of functioning. Scores range from 0 to 40. Higher scores indicate greater severity of symptoms.
Time Frame: Baseline to post-treatment (week 8); baseline to 2 months post-treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Present Centered Therapy (PCT)': The PCT is a form of individual therapy that is problem-oriented to improve current coping. It typically details of traumatic experiences. In this study, it is delivered individually in 8 weekly, 1 hour sessions to serve as an active, attention comparison arm. Sessions are unstructured and managed so that there is some engagement of the participant's emotional concerns with an emphasis on strengths and process encouragement rather than skills training. Three components of PCT include 1) developing a therapeutic relationship for social support, 2) focusing on current problems and problem solving, 3) and setting goals.
Arm/Group | Mantram Repetition Program (MRP) | Present Centered Therapy (PCT)'
Number analyzed (Participants) | 89 | 84
units on a scale
  Baseline | 25.01 (5.76) | 24.64 (5.64)
  Post-treatment | 18.01 (8.75) | 21.70 (6.53)
  2 months post-treatment | 17.61 (8.18) | 21.01 (6.87)
Statistical Analysis 1: Comparison: Mantram Repetition Program (MRP) vs Present Centered Therapy (PCT)'; This analysis is from baseline to post-treatment. Cronbach's alpha for this study was .78 at baseline; Test type: Superiority or Other; p < .006, Mixed Models Analysis — This p-value is based on a false discovery rate adjustment for multiple hypothesis testing
Statistical Analysis 2: Comparison: Mantram Repetition Program (MRP) vs Present Centered Therapy (PCT)'; This analysis is from baseline to 2 months post-treatment; Test type: Superiority or Other; p < .03, repeated measures — This p-value is based on a false discovery rate adjustment for multiple hypothesis testing

5. Secondary Outcome: Insomnia Severity Index (ISI)
Description: ISI is a widely used measure of insomnia with well-established reliability and validity. It consists of seven items, three of which assess severity of insomnia (i.e., degree of difficulty falling asleep, staying asleep, and waking too early). The remaining questions tap satisfaction with sleep pattern, effect of sleep on daytime and social functioning, and concern about current sleep difficulties. Both categorical and continuous measures of sleep difficulties can be assessed. Items are rated on a 0-4 Likert scale with higher scores meaning greater insomnia. Total scores range from 0-28. Original results were interpreted as 0-7 = no clinically significant insomnia, 8-14 = sub-threshold insomnia, 15-21 = moderately severe clinical insomnia and 21-28 = severe clinical insomnia. Later recommendations for a clinical, not community sample, are a cut-off of 11 points.
Time Frame: Baseline to post-treatment (week 8); baseline to 2 months post-treatment.
Population: Intent to treat analysis included 89 MRP and 84 PCT participants. Completers at post-treatment included 70 MRP and 72 PCT participants. Completers at 2-months follow up included 65 MRP and 71 PCT participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Present Centered Therapy: The PCT is a form of individual therapy that is problem-oriented to improve current coping. It typically details of traumatic experiences. In this study, it is delivered individually in 8 weekly, 1 hour sessions to serve as an active, attention comparison arm. Sessions are unstructured and managed so that there is some engagement of the participant's emotional concerns with an emphasis on strengths and process encouragement rather than skills training. Three components of PCT include 1) developing a therapeutic relationship for social support, 2) focusing on current problems and problem solving, 3) and setting goals.
Arm/Group | Mantram Repetition Program (MRP) | Present Centered Therapy
Number analyzed (Participants) | 89 | 84
units on a scale
  Baseline | 18.33 (6.59) | 16.34 (6.59)
  Post-treatment | 14.22 (7.47) | 16.62 (6.57)
  2 months post-treatment | 12.73 (7.90) | 15.92 (6.97)
Statistical Analysis 1: Comparison: Mantram Repetition Program (MRP) vs Present Centered Therapy; This analysis is from baseline to post-treatment. Cronbach's alpha for this study was .89 at baseline; Test type: Superiority or Other; p < 0.0008, repeated measures — This p-value is based on a false discovery rate adjustment for multiple hypothesis testing
Statistical Analysis 2: Comparison: Mantram Repetition Program (MRP) vs Present Centered Therapy; This analysis is from baseline to 2 months post-treatment; Test type: Superiority or Other; p < 0.006, Wilcoxon (Mann-Whitney) — This p-value is based on a false discovery rate adjustment for multiple hypothesis testing

6. Secondary Outcome: Patient Health Questionnaire (PHQ-9) for Depression
Description: PHQ-9 is a 9-item depression screening tool based on the diagnostic criteria for major depressive disorder in the DSM-IV. Each item is rated from a 0 (not at all) to 3 (nearly every day) scale. Items are summed and total scores range from 0 to 27. Higher scores indicate worse depression. A score of 11 or more considered probable depression and 20 or more is considered severe depression. It is well-validated and widely-used in medical settings such as primary care. The PHQ-9 includes the two major symptom domains characteristic of depression: affective and somatic symptoms.
Time Frame: Baseline to post-treatment (week 8); Baseline to 2-months post-treatment.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mantram Repetition Program (MRP) | Present Centered Therapy (PCT)
Number analyzed (Participants) | 89 | 84
units on a scale
  Baseline | 15.42 (5.89) | 15.15 (5.56)
  Post-treatment | 10.68 (6.19) | 12.81 (5.38)
  2 months post-treatment | 10.57 (6.37) | 12.18 (6.12)
Statistical Analysis 1: Comparison: Mantram Repetition Program (MRP) vs Present Centered Therapy (PCT); This analysis is from baseline to post-treatment. Cronbach's alpha for total score in this study was .86 at baseline; Test type: Superiority or Other; p < 0.10, Mixed Models Analysis — This p-value is based on a false discovery rate adjustment for multiple hypothesis testing. Raw p-value was <0.02
Statistical Analysis 2: Comparison: Mantram Repetition Program (MRP) vs Present Centered Therapy (PCT); This analysis is from baseline to post-treatment; Test type: Superiority or Other; p < 0.49, Mixed Models Analysis — This p-value is based on a false discovery rate adjustment for multiple hypothesis testing

7. Secondary Outcome: Spielberger State Anger Inventory-Short Form
Description: Spielberger State Anger Inventory-Short Form is a 10-item questionnaire with 4-point Likert scale to measure anger as an emotional state. Scores range from 10 to 40 with higher scores indicating more anger. Concurrent validity has been supported by correlations with measures of hostility, neuroticism, and anxiety. Internal consistency reliability has been reported as good to excellent.
Time Frame: Baseline to post-treatment (week 8); baseline to 2-months post-treatment.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 1: Mantram Repetition Program (MRP): The MRP teaches three portable, mindfulness strategies to train attention and manage symptoms: 1) Mantram (sacred word) Repetition, 2) Slowing Down, and 3) One-Pointed Attention. These tools are presented as working together synergistically and cumulatively, over time, to interrupt negative thoughts, behaviors, and emotional states such as anger, rage, irritability and impatience. Participants choose their own words or phrases and are encouraged to practice repeating a mantram at any time or place. In this study, MRP is delivered individually in eight weekly, 1-hour sessions, using a standardized manual, instructor guide, and homework assignments for experiential learning.
- Arm 2: Present Centered Therapy (PCT): The PCT is a form of individual therapy that is problem-oriented to improve current coping. It typically details of traumatic experiences. In this study, it is delivered individually in 8 weekly, 1 hour sessions to serve as an active, attention comparison arm. Sessions are unstructured and managed so that there is some engagement of the participant's emotional concerns with an emphasis on strengths and process encouragement rather than skills training. Three components of PCT include 1) developing a therapeutic relationship for social support, 2) focusing on current problems and problem solving, 3) and setting goals.
Arm/Group | Arm 1: Mantram Repetition Program (MRP) | Arm 2: Present Centered Therapy (PCT)
Number analyzed (Participants) | 89 | 84
units on a scale
  Baseline | 23.43 (9.78) | 12.00 (10.19)
  Post-treatment | 21.21 (8.58) | 22.20 (10.08)
  2 months post-treatment | 21.22 (9.18) | 21.27 (8.12)
Statistical Analysis 1: Comparison: Arm 1: Mantram Repetition Program (MRP) vs Arm 2: Present Centered Therapy (PCT); This analysis is from baseline to post-treatment. Cronbach's alpha for this study was .96 at baseline; Test type: Superiority or Other; p < 0.78, Mixed Models Analysis — This p-value is based on a false discovery rate adjustment for multiple hypothesis testing
Statistical Analysis 2: Comparison: Arm 1: Mantram Repetition Program (MRP) vs Arm 2: Present Centered Therapy (PCT); This analysis is from baseline to 2-months post-treatment; Test type: Superiority or Other; p < 0.99, Mixed Models Analysis — This p-value is based on a false discovery rate adjustment for multiple hypothesis testing

8. Primary Outcome: PTSD Checklist-Military Version [Diagnostic and Statistical Manual (DSM) IV-TR Version]
Description: PCL-M: PTSD Checklist-Military version (PCL-M) is a 17-item self-report screening instrument for PTSD symptoms related to military trauma. Items are scored on a 1 (not at all bothersome) to 5 (extremely bothersome) Likert scale. Total scores range from 17 to 85. Higher scores indicate greater symptom bothersomeness. A score of > 50 can suggest PTSD Test-retest reliability is high (r = 0.96) and validity is adequate, with a Kappa of 0.64 agreement for PTSD diagnosis compared to the Structured Clinical Interview for DSM-IV.
Time Frame: Baseline to post-treatment (week 8); Baseline to 2-months post-treatment.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mantram Repetition Program (MRP) | Present Centered Therapy (PCT)
Number analyzed (Participants) | 89 | 84
units on a scale
  Baseline | 59.23 (12.09) | 57.57 (11.56)
  Post-treatment | 45.32 (15.27) | 50.20 (13.92)
  2-months Post-treatment | 44.74 (14.58) | 48.42 (14.91)
Statistical Analysis 1: Comparison: Mantram Repetition Program (MRP) vs Present Centered Therapy (PCT); This analysis was from baseline to post-treatment. Cronbach's alpha for this study was .92 at baseline; Test type: Superiority or Other; p < 0.04, Mixed Models Analysis — This p-value is based on a false discovery rate adjustment for multiple hypothesis testing
Statistical Analysis 2: Comparison: Mantram Repetition Program (MRP) vs Present Centered Therapy (PCT); This analysis is from baseline to 2-months post-treatment; Test type: Superiority or Other; p < 0.25, Mixed Models Analysis — This p-value is based on a false discovery rate adjustment for multiple hypothesis testing

9. Secondary Outcome: Spielberger Trait Anger Inventory-Short Form
Description: Spielberger Trait Anger Inventory-Short Form is a 10-item questionnaire with 4-point Likert scale used to measure anger as a personality trait. Scores range from 10 to 40 with higher scores indicating more trait anger. Concurrent validity has been supported by correlations with measures of hostility, neuroticism, and anxiety. Internal consistency reliability has been reported as good to excellent.
Time Frame: Baseline to post-treatment (week 8); baseline to 2-months post-treatment.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Mantram Repetition Program (MRP) | Arm 2: Present Centered Therapy (PCT)
Number analyzed (Participants) | 89 | 84
units on a scale
  Baseline | 22.34 (7.16) | 21.89 (6.07)
  Post-treatment | 20.90 (6.95) | 10.37 (6.23)
  2-months post-treatment | 19.53 (6.81) | 18.62 (5.64)
Statistical Analysis 1: Comparison: Arm 1: Mantram Repetition Program (MRP) vs Arm 2: Present Centered Therapy (PCT); This analysis is from baseline to post-treatment. Cronbach's alpha for this study was .89 at baseline; Test type: Superiority or Other; p < 0.99, Mixed Models Analysis — This p-value is based on a false discovery rate adjustment for multiple hypothesis testing
Statistical Analysis 2: Comparison: Arm 1: Mantram Repetition Program (MRP) vs Arm 2: Present Centered Therapy (PCT); This analysis is from baseline to 2-months post-treatment; Test type: Superiority or Other; p < 0.94, Mixed Models Analysis — This p-value is based on a false discovery rate adjustment for multiple hypothesis testing

10. Secondary Outcome: Functional Assessment of Chronic Illness Therapy-Spiritual Wellbeing Scale-Expanded (FACIT-SpEx)
Description: The FACIT-SpEx was developed to assess spiritual components (e.g., harmony, meaning, purpose in life, peacefulness, faith/assurance) of quality of life using 23 items rated on a 5-point Likert scale from 0 (not at all) to 4 (very much). Total scores range from 0 to 92. Higher scores indicating greater spiritual well-being. Validity has been demonstrated by significant Pearson correlations between measures of quality of life, mood, and religious growth. It has demonstrated internal consistency reliability.
Time Frame: Baseline to post-treatment (week 8); baseline to 2-months post-treatment.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mantram Repetition Program (MRP) | Present Centered Therapy (PCT)
Number analyzed (Participants) | 89 | 84
units on a scale
  Baseline | 43.69 (17.84) | 44.74 (19.39)
  Post-treatment | 50.41 (17.24) | 46.28 (16.47)
  2 months Post-treatment | 50.95 (18.26) | 47.80 (19.42)
Statistical Analysis 1: Comparison: Mantram Repetition Program (MRP) vs Present Centered Therapy (PCT); This analysis is from baseline to post-treatment. Cronbach's alpha for this study was .88 at baseline; Test type: Superiority or Other; p < 0.12, Mixed Models Analysis — This p-value is based on a false discovery rate adjustment for multiple hypothesis testing
Statistical Analysis 2: Comparison: Mantram Repetition Program (MRP) vs Present Centered Therapy (PCT); This analysis is from baseline to 2-months post-treatment; Test type: Superiority or Other; p < 0.49, Mixed Models Analysis — This p-value is based on a false discovery rate adjustment for multiple hypothesis testing

11. Secondary Outcome: Five Facet Mindfulness Questionnaire (FFMQ)
Description: FFMQ a 39-item scale that measures five components of mindfulness: observing; describing; acting with awareness; non-judging of inner experience; and non-reactivity to inner experience. Each subscale contains either 7 or 8 items that are rated on a 1 (never or very rarely true) to 5 (very often or always true) Likert scale. Items are randomly reversed scored and higher scores represent greater levels of mindfulness. Total scores range from 39 to 195.
Time Frame: Baseline to post-treatment (week 8); baseline to 2-months follow-up.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Present Centered Therapy (PCT): The PCIT is a form of individual therapy that is problem-oriented to improve current coping. It typically details of traumatic experiences. In this study, it is delivered individually in 8 weekly, 1 hour sessions to serve as an active, attention comparison arm. Sessions are unstructured and managed so that there is some engagement of the participant's emotional concerns with an emphasis on strengths and process encouragement rather than skills training. Three components of PCT include 1) developing a therapeutic relationship for social support, 2) focusing on current problems and problem solving, 3) and setting goals.
Arm/Group | Arm 1: Mantram Repetition Program (MRP) | Present Centered Therapy (PCT)
Number analyzed (Participants) | 89 | 84
units on a scale
  Baseline | 121.34 (20.30) | 118.39 (17.33)
  Post-treatment | 121.29 (20.64) | 116.75 (19.56)
  2 months Post-treatment | 120.43 (21.40) | 119.00 (19.68)
Statistical Analysis 1: Comparison: Arm 1: Mantram Repetition Program (MRP) vs Present Centered Therapy (PCT); This analysis is from baseline to post-treatment. Cronbach's alpha for total score was .89 at baseline; Test type: Superiority or Other; p < 0.59, Mixed Models Analysis — This p-value is based on a false discovery rate adjustment for multiple hypothesis testing
Statistical Analysis 2: Comparison: Arm 1: Mantram Repetition Program (MRP) vs Present Centered Therapy (PCT); This analysis is from baseline to 2-months post-treatment; Test type: Superiority or Other; p < 0.10, Mixed Models Analysis — This p-value is based on a false discovery rate adjustment for multiple hypothesis testing; Mixed-effects, repeated measures models adjusting for demographic factors were implemented

ADVERSE EVENTS:
Time Frame: For 2 years of the study during active recruitment, enrollment, and study participation.
Arm/Group | Mantram Repetition Program (MRP) | Present Centered Therapy (PCT)
Serious Adverse Events (participants affected / at risk) | 1/89 | 3/84
Other Adverse Events (participants affected / at risk) | 0/89 | 0/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mantram Repetition Program (MRP) (N=89) | Present Centered Therapy (PCT) (N=84)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0) — Participant ran out of his prescription meds to treat depression. He went to the emergency room and was admitted to the hospital with a diagnosis of Depression Psychosis-Unspecified. He withdrew from the study.
Hospitalization for detoxification (Psychiatric disorders) | 0 (0) | 1 (1) — Participant was enrolled in study as clean and sober but relapsed. He was admitted to in-patient detoxification for substance abuse and follow-up after care. He remained in the research study.
Hospitalization for detoxification. (Psychiatric disorders) | 0 (0) | 1 (1) — Participant met study criteria upon enrollment, but had a relapse of substance abuse and was admitted to hospital for treatment. After detoxification, participant continued in the study.
Hospitalization for detoxification. (Psychiatric disorders) | 0 (0) | 1 (1) — Participant started using alcohol after 4 months of sobriety. He sought inpatient treatment and completed detoxification with follow-up. Participant remained in the study.

LIMITATIONS AND CAVEATS:
Study was to provide interventions for both conditions (MRP and PCT) in "group" format. Due to poor recruitment and after approval from Data Monitoring Committee, the study protocol was changed to provide both interventions in "individual" format.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes